CLINICAL TRIAL: NCT03338907
Title: Anesthesia vs Aviation: Does Added Carbon Dioxide in Normobaric Hypoxia Have the Same Effect on Cerebral Oxygenation as in Hypobaric Hypoxia?
Brief Title: CO2 (Carbon Dioxide) - Cerebral Oxygenation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-01790
Record Dates: First submitted 2017-10-30; First posted 2017-11-09 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Hypoxia, Brain
Keywords: cerebral hypoxia; CO2; cerebral perfusion; hypoxia
MeSH Terms: conditions — Hypoxia, Brain; Hypoxia

STUDY DESIGN:
Intervention Model Description: Controlled, randomized, single blind, crossover
Who Masked: Participant
Masking Description: The sequence whether the IMP or the comparator is applied first will be randomly assigned using the web-based randomizer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxycarbon (5% CO2 + 95% O2) (Experimental): Patients will be mechanical ventilated with Oxycarbon (5%CO2 +95% O2) after normocapnia is reached until FeO2 is stable for at least 1 min ≥ 80%. At timepoint 1 immediately prior apnea NIRS and vital parameters will be registered and an bloodsample will be drawn.
  Interventions: Drug: Oxycarbon (5% CO2+ 95% O2)
- Control (95% O2) (Placebo Comparator): Same procedure as arm "active comparator"
  Interventions: Drug: Oxycarbon (5% CO2+ 95% O2)

INTERVENTIONS:
Drug: Oxycarbon (5% CO2+ 95% O2) — Oxycarbon will be administered by mechanical ventilation

SUMMARY:
Several projects in high altitude research in environments with a low oxygen partial pressure (hypobaric hypoxia) leading to hypoxemia showed, that cerebral perfusion and cerebral performance could be improved by adding C02 (cabon dioxide).

The investigators hypothesize that adding 5% C02 to 02 (Oxygen) also under normobaric conditions increases the time until a significant cerebral hyopxia is measured by near infrared spectroscopy (NIRS) compared to the administration of 95% 02.

lf this hypothesis proves to be true, this approach might be used in situations in which individuals are prone to cerebral hypoxia. In bariatric surgery, patients that experience an apnea phase are more prone to (cerebral) hypoxia due to the fact, that they have a higher body mass index (BMI) leading to a reduced functional residual capacity (FRC), which serves as the oxygen reserve in the body.

DETAILED DESCRIPTION:
On the day of surgery patients will be randomized. After induction of anesthesia and endotracheal intubation patients will be managed by the study team to perform the intervention and the measurements.

According to randomization, investigational medical product (IMP) or comparator will be administrated by ventilator 1/ventilator 2.

At time point 1 apnea will be performed by disconnecting the ventilator from the endotracheal tube until the NIRS value has dropped by 20% from baseline. After that, re-ventilation will be resumed immediately, until parameters have returned to baseline.

During apnea time NIRS and vital signs will be recorded permanently, blood samples will be drawn at definite time points.

Application of IMP (or comparator) will be performed in this cross-over study design in the same manner after the baseline level is reached again.

At the end of the study procedure, after the baseline level of end-expiratory CO2 is reached again, patient will be taken over by the clinical anesthesia team and surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are designated for bariatric surgery at the University Hospital Zurich (USZ)
* Informed Consent as documented by signature
* BMI >35 kg/m2

Exclusion Criteria:

* Severe end-organ damage: chronic obstuctive pulmonary disease (COPD) GOLD (cassification) III and IV, known hepatic insufficiency or elevated liver enzymes, renal creatinine clearance <30ml/min
* Severe cardiovascular disease (NYHA classification III and IV)
* Known pulmonary Hypertension
* Cerebrovascular disease
* Pregnancy and lactation
* Cardiac dysrhythmias
* acidosis, chronic pulmonary disease
* Known or suspected non-compliance, drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Time to decrease of tissue oxygenation index by 20 % | 1 Day
  Parameter will be measured by NIRS

SECONDARY OUTCOMES:
PaO2 (Oxygen partial pressure) | 1 Day
  Parametere will be measured by arterial bloodgas
SpO2 (oxygen saturation) | 1 Day
  Parametere will be measured by arterial bloodgas
PCO2 ( partial pressure of carbon) | 1Day
  Parametere will be measured by arterial bloodgas

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schläpfer, MD, M.Sc., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Ist not planned to share data with other researchers

REFERENCES:
- [Background] Kety SS, Schmidt CF. THE EFFECTS OF ALTERED ARTERIAL TENSIONS OF CARBON DIOXIDE AND OXYGEN ON CEREBRAL BLOOD FLOW AND CEREBRAL OXYGEN CONSUMPTION OF NORMAL YOUNG MEN. J Clin Invest. 1948 Jul;27(4):484-92. doi: 10.1172/JCI101995. No abstract available. PMID 16695569
- [Background] Karl AA, McMillan GR, Ward SL, Kissen AT, Souder ME. Effects of increased ambient CO2 on brain tissue oxygenation and performance in the hypoxic rhesus. Aviat Space Environ Med. 1978 Aug;49(8):984-9. PMID 98161
- [Background] Brzecka A. Role of hypercapnia in brain oxygenation in sleep-disordered breathing. Acta Neurobiol Exp (Wars). 2007;67(2):197-206. doi: 10.55782/ane-2007-1648. PMID 17691228
- [Background] Kronenberg RS, Drage CW. Attenuation of the ventilatory and heart rate responses to hypoxia and hypercapnia with aging in normal men. J Clin Invest. 1973 Aug;52(8):1812-9. doi: 10.1172/JCI107363. PMID 4719663
- [Background] Hannay DR, Maddox EJ. Symptom prevalence and referral behaviour in Glasgow. Soc Sci Med (1967). 1976 Mar-Apr;10(3-4):185-9. doi: 10.1016/0037-7856(76)90046-9. No abstract available. PMID 968505
- [Background] Ainslie PN, Poulin MJ. Ventilatory, cerebrovascular, and cardiovascular interactions in acute hypoxia: regulation by carbon dioxide. J Appl Physiol (1985). 2004 Jul;97(1):149-59. doi: 10.1152/japplphysiol.01385.2003. Epub 2004 Mar 5. PMID 15004003